CLINICAL TRIAL: NCT00298181
Title: Controlled, Randomized, Prospective, Double-Blind, Multicenter, Phase I/II, Dose-Escalation Study of the Safety, PK, and Efficacy of YSPSL for Prevention of Delayed Graft Function in Patients Undergoing Cadaveric Kidney Transplantation
Brief Title: YSPSL for Prevention of Delayed Graft Function Part A
Status: Completed | Type: Observational
Sponsor: Y's Therapeutics, Inc. (Industry)
Responsible Party: Stefan Hemmerich, PhD, RAC, Y's Therapeutics Inc.
Other Study IDs: YSPSL-0001-PF Part A
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: Delayed Graft Function
MeSH Terms: conditions — Delayed Graft Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: YSPSL — YSPSL administered intravenously (IV) as a single bolus infusion open-label at 0.07, 0.22, 0.7 or 2.2 mg/kg
  Other Names: rPSGL-Ig; recombinant P-selectin glycoprotein ligand-Ig

SUMMARY:
Selectins have been implicated in the pathogenesis of ischemia/reperfusion (I/R)-induced kidney injury and resultant DGF. PSGL-1 is a ligand for P-, E-, and L-selectin. It has been reported that that YSPSL (rPSGL-Ig) blocks P-selectin and, to a lesser degree, E- and L-selectin. Both sPSGL-1 and YSPSL (rPSGL-Ig) have been shown in animal models to reduce both cytokines and tissue damage associated with ischemia reperfusion and to improve renal function post-transplant. Therefore, the current phase I/II clinical study is designed to assess the safety and efficacy of YSPSL (rPSGL-Ig) in preventing DGF in patients undergoing cadaveric kidney transplants and to determine a dose for future pivotal studies.

DETAILED DESCRIPTION:
This will be a multicenter, single-dose, dose-escalation study. The study will be in 2 parts: the first, Part A, will be an open label evaluation of single doses of four dose cohorts and the second, Part B will be a randomized, double-blind, placebo-controlled, single-dose, dose-escalation study of two dose cohorts. Patients who are undergoing cadaveric kidney transplantation and are at risk for development of DGF, based upon known risk factors, will be eligible to participate in the study. A maximum of 24 patients will be enrolled in Part A of the study. 60 patients will be enrolled in Part B.

ELIGIBILITY:
Inclusion Criteria:

* primary cadaver renal transplants Other inclusion criteria delineated in protocol

Exclusion Criteria:

* Full criteria delineated in protocol Patient has a planned transplant of a donor kidney from a non-heartbeating donor; Patient has a planned transplant of kidneys that are implanted en bloc (dual kidney transplant) or from donors <6 years of age; Patient has a planned transplant of a kidney from a donor who has received investigational therapies designed to reduce the impact of ischemia/reperfusion (I/R) injury, DGF, or other donor-related immune events; Patient is planned to receive a living donor kidney; or Patient is planned to receive an ABO-incompatible donor kidney.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-10; Primary Completion 2006-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
delayed graft function post transplant | 6 months

SECONDARY OUTCOMES:
renal function parameters through 6 months post transplant | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Hemmerich, PhD, Study Director — Y's Therapeutics, Inc.
Locations (10):
- United States (10):
  - Dumont-UCLA Transplant Center, Los Angeles, California
  - California Pacific Medical Center Department of Transplantation, San Francisco, California
  - Lifelink Foundation, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Westchester Medical Center, New York Medical College, Hawthorne, New York
  - University of Cincinnati, Department of Internal Medicine, Cincinnati, Ohio
  - Methodist Healthcare University Hospital, Memphis, Tennessee
  - Baylor University Medical Center Transplantation Services, Dallas, Texas
  - University of Texas, Organ Transplantation, Houston, Texas

REFERENCES:
- [Derived] Gaber AO, Mulgaonkar S, Kahan BD, Woodle ES, Alloway R, Bajjoka I, Jensik S, Klintmalm GB, Patton PR, Wiseman A, Lipshutz G, Kupiec-Weglinski J, Gaber LW, Katz E, Irish W, Squiers EC, Hemmerich S. YSPSL (rPSGL-Ig) for improvement of early renal allograft function: a double-blind, placebo-controlled, multi-center Phase IIa study. Clin Transplant. 2011 Jul-Aug;25(4):523-33. doi: 10.1111/j.1399-0012.2010.01295.x. Epub 2010 Jun 22. PMID 20573162